CLINICAL TRIAL: NCT01993082
Title: The Effects of Exercise and Life Stress on Telomere Maintenance and Cardiovascular Disease Risk
Brief Title: Fitness, Cellular Aging, and Caregiver Stress Study
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R00HL109247-03 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-25 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Aging; Stress; Disease Risk
Keywords: Caregivers; Telomerase; Telomere Length; Psychological Stress; Cardiovascular Risk; Exercise
MeSH Terms: conditions — Stress, Psychological; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Training Intervention (Experimental): For 24 weeks, subjects randomized into the aerobic training group will be asked to increase their physical activity level to meet the Centers for Disease Control and Prevention recommendations for physical activity of 150 minutes per week of moderate activity.
  A first visit with a fitness coach support provider, followed by weekly coaching texts and phone calls, will provide the framework for the activities in which participants should engage.
  Interventions: Behavioral: Aerobic Training Intervention
- Activity Maintenance Group (No Intervention): Participants randomized into the waitlist control group receive no aerobic training. Wait-list control participants will receive monthly check-in phone calls to establish that they have not significantly increased activity engagement. Participants in this group will receive a free gym membership at the end of the study, monthly phone calls with a fitness coach support provider for 6 months, and 2 coaching text messages per week.

INTERVENTIONS:
Behavioral: Aerobic Training Intervention — For 24 weeks, subjects randomized into the aerobic training group will be asked to increase their physical activity level to meet the Centers for Disease Control and Prevention recommendations for physical activity of 150 minutes per week of moderate activity.
  A first visit with a fitness coach support provider, followed by weekly coaching texts and phone calls, will provide the framework for the activities in which participants should engage.
  Arms: Aerobic Training Intervention

SUMMARY:
The purpose of this study is to determine whether an aerobic training intervention will alter markers of immune cell aging, improve exercise capacity and blood pressure and decrease psychological distress over 24 weeks in 32 caregivers compared to 32 age-matched wait list control caregivers.

DETAILED DESCRIPTION:
The investigators will prospectively examine whether an aerobic training intervention will alter markers of immune cell aging (i.e. increase telomerase activity in peripheral blood mononuclear cells, telomere length in peripheral blood mononuclear cells and leukocytes, mitochondrial function, epigenetic profiles, and mRNA expression), improve exercise capacity and blood pressure, and decrease psychological distress over 24 weeks in 32 caregivers compared to 32 age-matched wait list control caregivers. Our sample will be comprised of caregivers who provide unpaid care for a family member diagnosed with Alzheimer's disease or other dementia. Participants in the study will be highly stressed and inactive male and female caregivers of family members with Alzheimer's disease or other dementia. All eligible participants will complete one week of ecological momentary assessments (EMA) to examine whether (1) previously unfit, high-stressed caregivers benefit psychologically from becoming active, (2) this benefit is derived through changes in how caregivers react to and recover from stressful events, and (3) whether these salubrious psychological effects mediate changes in biological outcomes (e.g., cellular aging). Next, participants will participate in a one-week run-in period of stretching 30 minutes on 4 separate days prior to randomization to guarantee that the investigators are randomizing well-informed participants that are willing and able to complete the expected exercise. Next, participants are randomized into the aerobic exercise or wait list control arm. In the 24th week of the study, participants complete a second week of the EMAs sub-study, and return after week 24 for a final blood draw.

Research study assessments consist of self-report questionnaires, body composition, physical performance and fitness tests, and a fasting blood draw. The follow-up visit, 24 weeks later, consists of a repeat of the same morning health visit.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-75
* Men and Women (women must be post-menopausal)
* Body Mass Index must be below 40 (to exclude for extreme obesity, which can confound outcomes)
* Must be a first or second degree family member providing unpaid caregiving for an adult relative with Alzheimer's disease or other dementias of longer than 6 months since diagnosis.
* Must report providing care for 10 or more hours per week.
* Perceived stress ≥ 15 for adults 65 and older; Perceived stress ≥ 18 for adults aged 50-64. (0.5 standard deviation above national average for adults)
* Do not meet Center for Disease Control recommendations for exercise (150 minutes per week of moderate activity levels or 75 minutes of vigorous)

Exclusion Criteria:

* Major Chronic Disease that interferes with activity levels as advised by a medical practitioner (Autoimmune disorders; severe asthma; lung disease - emphysema or chronic bronchitis; history of stroke, heart attack, cardiovascular disease, epilepsy, or brain injury)
* Heart attack in the past 6 months or repeated experience of chest pain or pressure, and/or arrhythmia.
* Cancer that is not in remission. Those who underwent chemotherapy or radiation within the past 5 years will be excluded.
* Eating Disorders
* Current substance dependence that can interfere with activity engagement.
* Current Post Traumatic Stress Disorder
* Current or recent smoking status. We will exclude current smokers and past smokers (who quit within the past 5 years).
* Confounding medications- Oral Steroids containing prescription drugs use and any other drugs that might interfere with the outcome measures.
* Current major injuries
* Any physical impairment that prevent participation in moderate levels of physical activity (e.g. musculoskeletal problems, prosthesis)
* Inability to walk a block or climb stairs without chest pain, losing breath, or dizziness

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Telomerase in Peripheral Blood Mononuclear Cells | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in Telomerase in Peripheral Blood Mononuclear Cells at 24 weeks. Participants will provide blood samples at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study.

SECONDARY OUTCOMES:
Change in Cardiovascular Fitness | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in Cardiovascular Fitness at 24 weeks. Participants will participate in fitness testing (treadmill test and respiratory gas analysis/ V02 Peak) at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study.
Change in Diastolic and Systolic Blood Pressure | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in Change in Diastolic and Systolic Blood Pressure at 24 weeks. Study staff will measure blood pressure at participant's baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study.
Change in Psychological Well-being (general and daily) | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in Change in Psychological Well-being (general and daily) at 24 weeks. We will collect perceived stress, caregiving burden, depression measures, emotion regulation, marital satisfaction, rumination, anxiety, self-esteem, and other measures of psychological well-being and distress at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study. We will also have ecological momentary assessments six times a day for one week prior to the intervention and again in the final, 24th, week of the study to examine changes in stress sensitivity as a result of exercise.
Change in Telomere Length in Leukocyte/ Peripheral Blood Mononuclear Cells | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in Telomere Length in Leukocyte/ Peripheral Blood Mononuclear Cells at 24 weeks. Participants will provide blood samples at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study. We will measure telomere length pre- and post-intervention in Leukocyte and Peripheral Blood Mononuclear Cells.
Change in Mitochondrial Functioning (Enzyme Activity, DNA Copy Number) in Peripheral Blood Mononuclear Cells | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in Mitochondrial Functioning in Peripheral Blood Mononuclear Cells at 24 weeks. Participants will provide blood samples at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study.
Change in Epigenetic Aging Profiles | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in Epigenetic Aging Profiles (i.e. Methylation), at 24 weeks. Participants will provide blood samples at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study.
Change in mRNA expression | Measured at Week 0 (baseline) and Week 24
  Change from Baseline in mRNA expression, at 24 weeks. Participants will provide blood samples at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 24th week of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Epel, PhD, Principal Investigator — University of California, San Francisco; Samantha Schilf, BA, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States